CLINICAL TRIAL: NCT01918670
Title: A French Multi-centric Atrial Fibrillation Catheter Ablation Survey
Acronym: FrenchAF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinique Pasteur (Other)
Collaborators: University Hospital, Grenoble (Other); Nouvelle Clinique Nantaise, Nantes, France (Unknown); Hôpital Privé de Parly II - Le Chesnay (Other); Rennes University Hospital (Other); University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Serge Boveda, MD, Clinique Pasteur
Other Study IDs: FrenchAFAblationSurvey
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Observation of Outcome After Catheter Ablation of Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; relapse; stroke; death
MeSH Terms: conditions — Atrial Fibrillation; Recurrence; Stroke; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Pasteur
  Interventions: Procedure: catheter ablation of atrial fibrillation
- Grenoble
  Interventions: Procedure: catheter ablation of atrial fibrillation
- Nantes
  Interventions: Procedure: catheter ablation of atrial fibrillation
- Parly
  Interventions: Procedure: catheter ablation of atrial fibrillation
- Rennes
  Interventions: Procedure: catheter ablation of atrial fibrillation
- Rouen
  Interventions: Procedure: catheter ablation of atrial fibrillation

INTERVENTIONS:
Procedure: catheter ablation of atrial fibrillation — electric pulmonary vein disconnection

SUMMARY:
Atrial fibrillation is the most frequent sustained arrhythmia. Catheter ablation is a procedure that is currently used for the treatment of symptomatic atrial fibrillation patients.

We have organized a multi-centric national survey of catheter ablation of atrial fibrillation in order to have a feedback on the type of procedures being performed and the overall results (freedom of atrial fibrillation) over an average follow-up of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing catheter ablation of atrial fibrillation or left atrial flutter

Exclusion Criteria:

* patients undergoing catheter ablation of other types of arrhythmia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing catheter ablation in one of the registry centers
Sampling Method: Non-Probability Sample
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation relapse | starting 3 months after the procedure till an average of 18months follow-up
  Documentation of atrial fibrillation relapse (symptomatic or asymptomatic) after the first 3 months after the index procedure

SECONDARY OUTCOMES:
Early atrial fibrillation relapse | first 3 months
  Documented atrial fibrillation relapse (symptomatic or asymptomatic) in the first 3 months after the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pasteur, Toulouse, France